CLINICAL TRIAL: NCT05330507
Title: POWER: Prospective, Observational Study of Wellinks Effect on COPD Hospital Readmissions
Brief Title: Prospective, Observational Study of Wellinks Effect on COPD Hospital Readmissions
Acronym: POWER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Convexity Scientific Inc (Industry)
Collaborators: Hartford HealthCare (Other)
Responsible Party: Sponsor
Other Study IDs: WL-2022-01-HHC
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: COPD; Respiratory Tract Disease; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Lung Diseases
Keywords: Exacerbation; Discharge; Hospitalization; Readmission; Virtual Care; Digital Health; V1C
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wellinks Intervention: Following inpatient hospitalization for COPD exacerbation, participants will receive 16 weeks of access to Wellinks (i.e., connected spirometer and pulse oximeter, virtual respiratory therapist sessions with pulmonary rehabilitation, virtual health coaching sessions, mobile app access, COPD-related education). The 16-week period is comprised of a 30-day post-discharge program followed by a 12-week intensive period, which vary by frequency of contact with respiratory therapists/health coaches.
  Interventions: Other: Wellinks
- Matched Controls: A matched control dataset will be extracted from electronic medical records of the participating healthcare system. Participants will be matched on an index COPD-related hospitalization and other key factors, utilizing propensity score matching (i.e., number of COPD-related hospitalizations in prior year, severity of COPD, age).

INTERVENTIONS:
Other: Wellinks — 30-day post-discharge period: virtual respiratory therapist sessions twice per week with synchronous virtual pulmonary rehabilitation and educational materials; at-home use of connected spirometer and pulse oximeter; at-home use of mobile app.
  12-week intensive period: virtual health coaching sessions once every two weeks; asynchronous virtual pulmonary rehabilitation program; ongoing access to connected devices (spirometer and pulse oximeter) and mobile app.
  Groups: Wellinks Intervention

SUMMARY:
This prospective, observational study is designed to investigate clinical outcomes and collect patient feedback on the use of Wellinks, an integrated virtual chronic obstructive pulmonary disease (COPD) management solution, for patients recently discharged from the hospital due to an acute exacerbation of their COPD.

DETAILED DESCRIPTION:
Wellinks, an integrated virtual COPD management solution consists of a combination of health coaching, Bluetooth-connected devices, collection of patient-reported symptoms and medication use, and virtual pulmonary rehabilitation, all centralized by the use of a mobile-phone application (mobile app) downloaded onto a study participant's iOS (iPhone) or Android device. The clinical objectives of this study are to determine whether utilization of Wellinks can reduce the rate of hospital readmissions due to a COPD exacerbation for patients recently discharged from the hospital. The nonclinical objectives of this study are to describe the experience of study participants using Wellinks through the assessment of engagement with the components of Wellinks, as well as by participant-reported satisfaction and perceived value (e.g., willingness to pay). Qualitative feedback on the features and functionality of Wellinks will be solicited.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age with no upper age limit) 2. Any sex, race and ethnicity 3. COPD diagnosis 4. Current hospital admission or observation status resulting from exacerbation of COPD or generally including respiratory signs/symptoms indicative of difficulty breathing (e.g., need for oxygen or nebulized therapy, increased use of rescue medication) 4. Telephone (landline or mobile) and internet access 5. Access to a smartphone: iPhone 6S or later model, running iOS 14.0 or later; Android 6 or later model 6. Proficient in English language due to the availability of all study materials in the English language only 7. Living/staying in the United States throughout the study duration 8. Eligible to participate in asynchronous virtual pulmonary rehabilitation in the opinion of the investigator (e.g., patients determined to be ineligible to participate may include those with acute coronary syndrome for whom an exercise regimen is not advisable at present time) 9. Willing and able to comply with study requirements 10. Able to provide written informed consent

Exclusion Criteria:

1. Diagnosis of acute decompensated heart failure
2. Currently pregnant or planning to become pregnant during the study period
3. Life expectancy <17 weeks
4. Current participation in other interventional clinical trials
5. Current participation in a pulmonary rehabilitation program

7. Enrollment in an existing Wellinks program 8. Unable or unwilling to cooperate with remote assessments and engagement with Coaches 9. Unable to comply with the study procedures in the opinion of the investigator (e.g., unlikely to be compliant, unlikely to comprehend instructions or education provided)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with COPD hospitalized due to a COPD exacerbation are eligible for enrollment into the Wellinks intervention. Study participants are required to fulfill certain criteria for access to the internet and a smartphone. Key exclusion criteria are congestive heart failure for the potential risk to participation in virtual pulmonary rehabilitation, coincident SARS-CoV-2 infection due to the unknown impact on the post-discharge outcomes of COPD patients, and current participation in other interventional programs or active engagement in pulmonary rehabilitation. See complete list of eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Hospital readmission rate (all-cause) | 30-days post-discharge from index event
  Rate of all-cause hospital readmission
Hospital readmission rate (all-cause) | 60-days post-discharge from index event
  Rate of all-cause hospital readmission
Hospital readmission rate (all-cause) | 90-days post-discharge from index event
  Rate of all-cause hospital readmission
Hospital readmission rate (COPD-related) | 30-days post-discharge from index event
  Rate of COPD-related hospital readmission
Hospital readmission rate (COPD-related) | 60-days post-discharge from index event
  Rate of COPD-related hospital readmission
Hospital readmission rate (COPD-related) | 90-days post-discharge from index event
  Rate of COPD-related hospital readmission
COPD Assessment Test | Change from baseline to day 30 (end of post-discharge intervention phase) and to week 16 (end of study)
  Assess quality-of-life impact of COPD
Exercise capacity: 30-second sit-to-stand | Change from baseline to day 30 (end of post-discharge intervention phase) and to week 16 (end of study)
  Assess exercise capacity
Modified Medical Research Council Dyspnea Index (mMRC) | Change from baseline to day 30 (end of post-discharge intervention phase) and to week 16 (end of study)
  Assess shortness of breath and impact on daily activities

SECONDARY OUTCOMES:
Wellinks App Engagement | 16 weeks
  Frequency of use of the mobile app throughout the study period
Wellinks Device Engagement | 16 weeks
  Frequency of use of the connected devices throughout the study period
Wellinks Session Engagement | 16 weeks
  Participation rate in scheduled respiratory therapist and health coaching sessions
Patient Satisfaction (Net Promoter Score) | 16 weeks
  Net promoter score from asking, "How likely is it that you would recommend Wellinks to a friend or colleague?"

OTHER OUTCOMES:
Value Ranking of Wellinks Features | 16 weeks
  Value ranking of the various components of Wellinks

CONTACTS AND LOCATIONS:
Overall Officials: Syed Hadi, MD, Principal Investigator — Hartford HealthCare
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No